CLINICAL TRIAL: NCT02142842
Title: Phase I/II Study of Transplantation of Autologous Adipose Stem Cells and Activated Platelet Rich Plasma in Knee Osteoarthritis Treatment
Brief Title: Autologous Adipose Stem Cells and Platelet Rich Plasma Therapy for Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Science Ho Chi Minh City (Other)
Collaborators: GeneWorld Co., Ltd., Ho Chi Minh (Unknown); Van Hanh General Hospital (Other); 115 People's Hospital (Other Government)
Responsible Party: Principal Investigator, Phuc Van Pham, Laboratory of Stem Cell Research and Apllication, University of Science Ho Chi Minh City
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1438/QDBYT
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Knee Osteoarthritis
Keywords: Adipose stem cell; Platelet rich plasma; Knee Osteoarthritis; Injured cartilage
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Autologous stromal vascular fraction (SVF) and platelet rich plasma (PRP) will be injected into joints of 16 patients with grade 2, 3 radiographic OA severity with 16 patients as control.
  Interventions: Biological: Autologous adipose tissue stromal vascular fraction and platelet rich plasma

INTERVENTIONS:
Biological: Autologous adipose tissue stromal vascular fraction and platelet rich plasma

SUMMARY:
Adipose stem cells and platelet rich plasma can regenerate the injured cartilage.

DETAILED DESCRIPTION:
The proposed study is two centers, unblinded, non randomized, phase I/II trial in which the patients will be treated with a single dose of autologous stromal vascular cells (SVF) in combination with platelet rich plasma (PRP).

This study aimes to evaluate the clinical efficiency of autologous adipose tissue-derived MSC transplantation in patients with confirmed osteoarthritis at grade II and III. Adipose tissue is isolated from the belly, and used for extraction of the SVF. The SVF is mixed with activated platelet-rich plasma before injection. The clinical efficiencies are evaluated by the pain score (VAS), Lysholm score, and MRI findings. SVF is isolated from about 100 mL of adipose tissue, and PRP is prepared from 20 mL of peripheral blood. Total injection volume will be about 5-10 mL. The total number of SVF to be injected is 1.0 x 10(7) to 5 x 10(7).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and ability to understand the planned treatment.
* Idiopathic or secondary osteoarthritis of the knee with grade 2, 3 radiographic severity

Ability and willingness to undergo liposuction

Exclusion Criteria:

* Pregnant women or cognitively impaired adults.
* Presence of large meniscal tears ("bucket handle" tears), as detected by clinical examination or by magnetic resonance imaging.
* Inflammatory or postinfectious arthritis.
* More than 5 degrees of varus or valgus deformity.
* Kellgren Lawrence grade 4 osteoarthritis in two compartments (the medial or lateral compartments of the tibiofemoral joint or the patellofemoral compartment) in persons over 60 years of age.
* Intraarticular corticosteroid injection within the previous 3 months.
* A major neurologic deficit.
* Serious medical illness with a life expectancy of less than 1 year.
* Prior admission for substance abuse
* Body Mass Index (BMI) of 40 kg/m2 or greater
* Patient receiving experimental medication or participating in another clinical study within 30 days of signing the informed consent
* In the opinion of the investigator or the sponsor the patient is unsuitable for cellular therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 6 months

SECONDARY OUTCOMES:
Change from the baseline pain score (VAS) at 6 months | 6 months, 12 months, 18 months
Change from baseline Lysholm score at 6 months | 6 months, 12 months, 18 months
Change from baseline MRI assessment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Phuc V Pham, PhD, Study Director — Laboratory of Stem Cell Research and Application, University of Science, VNU-HCM, VN; Phuong TB Le, MSc, MD, Principal Investigator — Van Hanh Hospital, Ho Chi Minh city, VN; Phu D Nguyen, PhD, MD, Principal Investigator — 115 Hospital, HCM; Ho H La, MD, Principal Investigator — Van Hanh Hospital, Ho Chi Minh city, VN; Tung DX Tran, MSc, MD, Principal Investigator — Van Hanh Hospital, Ho Chi Minh city, VN
Locations (3):
- Vietnam (3):
  - 115 Hospital, Ho Chi Minh city, Ho Chi Minh City
  - Laboratory of Stem Cell Research and Application, University of Science, Vietnam National University, Ho Chi Minh, Ho Chi Minh City
  - Van Hanh Hospital, Ho Chi Minh city, VN, Ho Chi Minh City